CLINICAL TRIAL: NCT00049192
Title: A PHASE II STUDY OF G3139 (GENASENSE™, NSC # 683428 IND # 58842) + IMATINIB MESYLATE (GLEEVEC®, STI571) IN PATIENTS WITH IMATINIB-RESISTANT CHRONIC MYELOID LEUKEMIA
Brief Title: Oblimersen and Imatinib Mesylate in Treating Patients With Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02790; CALGB 10107; U10CA031946 (NIH)
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Chronic Phase Chronic Myelogenous Leukemia; Relapsing Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase | interventions — oblimersen; Imatinib Mesylate

ARMS (1):
- Treatment (oblimersen sodium, imatinib mesylate) (Experimental): Patients receive oblimersen IV continuously on days 1-10 and oral imatinib mesylate once or twice daily. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients without a hematologic response after 2 courses go off study. Patients with complete or partial response after 4 courses may continue to receive oral imatinib mesylate daily.
  Patients in cohort 2 receive an escalated dose of oblimersen; if well tolerated, subsequent cohorts receive oblimersen at the higher dose with the original dose of imatinib mesylate. If oblimersen is not well tolerated in cohort 2, subsequent cohorts receive the original dose of oblimersen with an escalated dose of imatinib mesylate. The first 6 patients accrued continue to receive the original dose (dose taken prior to study) of imatinib mesylate throughout the study.
  Interventions: Biological: oblimersen sodium; Drug: imatinib mesylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: oblimersen sodium — Given IV
  Other Names: augmerosen; G3139; G3139 bcl-2 antisense oligodeoxynucleotide; Genasense
Drug: imatinib mesylate — Given PO
  Other Names: CGP 57148; Gleevec; Glivec
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of combining oblimersen with imatinib mesylate in treating patients who have chronic myelogenous leukemia that has not responded to previous treatment with imatinib mesylate. Imatinib mesylate may stop the growth of cancer cells by blocking the enzymes necessary for cancer cell growth. Oblimersen may help imatinib mesylate kill more cancer cells by making cancer cells more sensitive to the drug.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the cytogenetic response rate of patients with CML who have had less than a complete hematologic response or less than major cytogenetic response to imatinib mesylate and who have been treated after two cycles of imatinib mesylate + G3139.

SECONDARY OBJECTIVES:

I. To estimate the hematologic, cytogenetic and molecular response rate and duration in patients diagnosed with CML who have been treated after two and four cycles of imatinib mesylate + G3139.

II. To estimate the toxicity of these two drugs given in combination in a cooperative group setting.

OUTLINE:

Patients receive oblimersen IV continuously on days 1-10 and oral imatinib mesylate once or twice daily. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients without a hematologic response after 2 courses go off study. Patients with complete or partial response after 4 courses may continue to receive oral imatinib mesylate daily.

Patients in cohort 2 receive an escalated dose of oblimersen; if well tolerated, subsequent cohorts receive oblimersen at the higher dose with the original dose of imatinib mesylate. If oblimersen is not well tolerated in cohort 2, subsequent cohorts receive the original dose of oblimersen with an escalated dose of imatinib mesylate. The first 6 patients accrued continue to receive the original dose (dose taken prior to study) of imatinib mesylate throughout the study.

Patients are followed monthly for 3 months and then every 3 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic myeloid leukemia (CML) in chronic phase; clonal cytogenetic evolution alone does not exclude patients
* Patients in whom a Philadelphia chromosome [t(9;22)] or a variant translocation is not detectable by cytogenetic studies are eligible if they meet one of the following criteria:

  * Polymerase chain reaction (PCR) positive fusion transcripts for BCR/ABL;
  * BCR/ABL translocation present by fluorescence in situ hybridization (FISH)
* Patients must have received prior therapy with imatinib mesylate (>= 400 mg/day for > 8 weeks without a complete hematologic response or >= 400 mg/day for > 6 months without a major cytogenetic response) and must not have evidence of progressive disease (accelerated or blast phases)
* Patients must have received a stable dose of imatinib mesylate >= 600 mg/day for at least 4 weeks without > grade 1 toxicities; the first six patients enrolled will be restricted to receiving an imatinib mesylate dose of 600 mg/day while on study
* No prior therapy with hydroxyurea, cytarabine, interferon, anagrelide, homoharringtonine, or any other investigational agent within 4 weeks of study enrollment
* Patients may not have received other antineoplastic medications (e.g., busulfan)
* No prior stem cell transplantation
* Patients must not require oral anticoagulant therapy
* Non-pregnant and non-nursing; treatment under this protocol would expose an unborn child to significant risks. Women and men of reproductive potential should agree to use an effective means of birth control throughout the duration of protocol treatment and for at least three months after the last dose of imatinib mesylate
* No other serious illnesses which would limit survival to < 2 years, or a psychiatric condition which would prevent compliance with treatment or informed consent
* No uncontrolled cardiovascular disease, diabetes, pulmonary disease, or infection, which in the opinion of the treating physician, would make this protocol treatment unreasonably hazardous for the patient
* Patients with a "currently active" second malignancy other than non-melanoma skin cancers are not eligible; patients are not considered to have a "currently active" malignancy if they have completed therapy and are considered by their physician to be at less than 30% risk of relapse within one year
* Bilirubin =< 2 mg/dL
* Creatinine =< 2 mg/dL
* AST =< 1.5 x Upper Limit of Normal
* PTT =< 1.5 x Upper limit of Normal
* BHCG Negative (if patient of childbearing potential)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2002-11; Primary Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Cytogenetic response rate in bone marrow | 42 days

SECONDARY OUTCOMES:
Hematologic response rate in peripheral blood | Up to 84 days
Cytogenetic response rates | Up to 84 days
Molecular response rates | Up to 84 days
Duration of response | Up to 5 years
Toxicities of concomitant treatment, reported using the NCI Common Toxicity Criteria version 2.0 | Up to 30 days after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Meir Wetzler, Principal Investigator — Cancer and Leukemia Group B
Locations (1):
- Cancer and Leukemia Group B, Chicago, Illinois, United States